CLINICAL TRIAL: NCT06896695
Title: Financial Compass: A Pilot Feasibility Study of a Novel Intervention to Identify and Address Financial Hardship Among Cancer Patients
Brief Title: A Financial Intervention (Financial Compass) to Identify and Address Financial Hardship Among Head and Neck Cancer Patients, Financial Compass Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I-4123124; NCI-2025-01528 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-4123124 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aim 1 (interview) (Other): Patients complete interviews on study for Financial Compass intervention development and refinement.
  Interventions: Other: Interview
- Aim 2 (discussion) (Other): Participants take part in a community advisory board and/or a health care delivery advisory board on study to discuss, develop and refine the Financial Compass intervention.
  Interventions: Other: Discussion
- Aim 3 Group I (Financial Compass intervention) (Experimental): Patients receive the Financial Compass intervention on study including a patient needs assessment, a tailored care pathway and weekly individualized navigation and support to access resources.
  Interventions: Other: Financial Navigation; Other: Survey Administration
- Aim 3 Group II (usual care) (Active Comparator): Patients receive usual care on study including medical consultations and supportive care.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Aim 3 Group II (usual care)
Other: Discussion — Ancillary studies
  Other Names: Discuss
  Arms: Aim 2 (discussion)
Other: Financial Navigation — Receive the Financial Compass intervention
  Other Names: Financial Navigation Program
  Arms: Aim 3 Group I (Financial Compass intervention)
Other: Interview — Ancillary studies
  Arms: Aim 1 (interview)
Other: Survey Administration — Ancillary studies
  Arms: Aim 3 Group I (Financial Compass intervention); Aim 3 Group II (usual care)

SUMMARY:
This clinical trial compares the effect a financial intervention, called Financial Compass, to usual care in identifying and addressing financial hardship in patients with head and neck cancer. Previous research has shown that head and neck cancer patients experiencing financial hardship have decreased overall and cancer specific survival. Using a financial intervention, Financial Compass, may be more effective than usual care in identifying and addressing financial hardship in patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine head and neck cancer patients' experiences with financial hardship to understand barriers across the socioeconomic spectrum and inform intervention refinement. (Aim 1) II. Apply community-engaged intervention mapping to tailor the Financial Compass intervention to address the needs and experiences of head and neck cancer patients. (Aim 2) III. Conduct a pilot randomized control trial of Financial Compass to assess feasibility, acceptability and preliminary efficacy among head and neck cancer patients. (Aim 3)

OUTLINE:

AIM 1: Patients complete interviews on study for Financial Compass intervention development and refinement.

AIM 2: Participants take part in a community advisory board and/or a health care delivery advisory board on study to discuss, develop and refine the Financial Compass intervention.

AIM 3: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive the Financial Compass intervention on study including a patient needs assessment, a tailored care pathway and weekly individualized navigation and support to access resources.

GROUP II: Patients receive usual care on study including medical consultations and supportive care.

After completion of study intervention, patients are followed up at week 12.

ELIGIBILITY:
Inclusion Criteria:

* They have been diagnosed with head and neck cancer
* Screen positive for financial hardship on the validated Comprehensive Score for Financial Toxicity (COST) measure
* Are able to participate in English or Spanish

Exclusion Criteria:

* Adults unable to complete the process of informed consent
* Adults whose primary language is not English or Spanish
* Individuals who are not yet adults (i.e., infants, children, teenagers)
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-02-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Cancer-related financial hardship (Aim 1) | Up to 2 years
  Will make significant conceptual contributions to the understanding of the experience of cancer-related financial hardship and differences in needs and barriers by income levels. Findings will make significant translational impact through identifying domains for intervention tailoring for the Financial Compass intervention. Qualitative data will be coded and analyzed. Will use thematic analysis to categorize and identify themes. Will use multiple coders to increase reliability. Any coding discrepancies will be discussed and resolved using a consensus approach. Qualitative data will be summarized.
Development of the Financial Compass intervention (Aim 2) | Up to 2 years
  Will use stage 1A of the National Institutes of Health Stage Model to further develop the Financial Compass intervention. Will use data from in-depth interviews and collaborative engagement of advisory boards to refine the final Financial Compass intervention package. Will complete the Financial Compass intervention package. Will use the Person, Extended Family, Neighborhood (PEN)-3 model to guide integration of stakeholder feedback into the final Financial Compass intervention package. Will prepare summaries of key findings from the in-depth interviews to review with advisory board members. Themes in advisory board member feedback will be categorized using the main constructs of PEN-3 model in a 3 x 3 table, including (1) perceptions, (2) enablers, and (3) nurturers.
Feasibility of the Financial Compass intervention (Aim 3) | Up to 12 weeks
  Will assess feasibility of the Financial Compass intervention among head and neck cancer patients. Will examine feasibility through demand (study enrollment rates, reasons for refusal), practicality (retention rates, engagement with intervention sessions/materials, reasons for study drop out), and acceptability (participant satisfaction with intervention materials and content). To assess acceptability, will administer the Acceptability of Intervention Measure (4 items), Intervention Appropriateness Measure (4 items) and Feasibility of Intervention Measure (4 items). The measures use a 5-point Likert scale where 1 = completely disagree and 5 = completely agree and have demonstrated strong psychometric properties. In the Financial Compass group, the measures will be summarized using the appropriate descriptive statistics, with estimates of enrollment and retention rates obtained with 90% confidence intervals.
Efficacy of the Financial Compass intervention (Aim 3) | Up to 12 weeks
  Will assess efficacy of the Financial Compass intervention among head and neck cancer patients. Will use the Comprehensive Score for Financial Toxicity (COST), an 11-item measure that captures participants' financial concerns. Will compare COST scores between groups using a one-sided t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States